CLINICAL TRIAL: NCT04305886
Title: Interprofessional Group Intervention to Promote Faculty Wellbeing and Engagement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Susan Hata, MD, Co- Investigator, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2018P000415
Record Dates: First submitted 2020-03-03; First posted 2020-03-12 (Actual); Last update posted 2020-03-12 (Actual); Status verified 2020-03

CONDITIONS: Burnout, Professional
MeSH Terms: conditions — Burnout, Professional

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Providers were placed in small groups and given the intervention of a discussion guide to facilitate discussion.
  Interventions: Other: Discussion Guide
- Control (No Intervention): Providers were placed in small groups and not given a discussion guide to facilitate discussion.

INTERVENTIONS:
Other: Discussion Guide — Written list of prompts to facilitate discussion
  Arms: Intervention

SUMMARY:
A randomized trial of an interprofessional intervention to reduce burnout and enhance professional engagement in physicians, certified nurse midwives, and nurse practitioners.

DETAILED DESCRIPTION:
To test the hypothesis that an intervention involving self-facilitated interprofessional group meetings would result in improvement in wellbeing and to determine whether use of a written curriculum provided increased benefit, the following study is conducted:

Practicing clinical faculty in the Department of Obstetrics and Gynecology at the Massachusetts General Hospital were recruited to participate in three monthly small groups over dinner. Participants were randomized to a control group, which met without any specified guidelines for discussion content, or to receive an intervention which consisted of a one-page discussion guide addressing themes relevant to challenges in the healthcare environment: reframing challenging patient interactions; embracing uncertainty in work; and coping with errors, near misses, and bad outcomes. Outcomes included burnout, empowerment and engagement in work, stress from uncertainty assessed using validated metrics, and perception of of collegiality and community.

All participants were also offered the option of participating in evaluation of biomarkers. To test the hypothesis that an increased sense of bonding and relational connection, and reduced stress levels would be reflected by changes in hormone levels during the meeting and over the course of the study. Faculty who opted into this portion of the study gave the following samples:

Urine Oxytocin before and after the first and third group meetings Salivary Oxytocin before and after the first and third group meetings Salivary Cortisol before and after the first and third group meetings Hair Cortisol at the beginning of the study and at the end of the study (a roughly three month interval).

An optional focus group was conducted after the three monthly sessions.

All participants signed a consent form prior to participating in the study.

ELIGIBILITY:
Inclusion Criteria:

* Physican in the Department of Obstetrics and Gynecology at Massachusetts General Hospital
* Nurse Practitioner in the Department of Obstetrics and Gynecology at Massachusetts General Hospital
* Certified Nurse Midwife in the Department of Obstetrics and Gynecology at Massachusetts General Hospital

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2018-09-30 (Actual); Study Completion 2018-09-30 (Actual)

PRIMARY OUTCOMES:
Burnout | Change over the three month study period. Baseline measurement and immediately after final intervention.
  Change from baseline in 2 item Maslach Burnout Inventory scores before and after the intervention.
  Minimum score: 2; Maximum score: 14 Higher score = more burnt out (worse outcome)
Stress from Uncertainty | Change over the three month study period. Baseline measurement and immediately after final intervention.
  Change in scores on Physician Response to Uncertainty Scale before and after intervention Minimum score: 6; Maximum score: 90 Higher score = increased stress due to uncertainty (worse outcome)
Work Engagement | Change over the three month study period. Baseline measurement and immediately after final intervention.
  Change in scores on Utrecht Work Engagement Scale before and after intervention Minimum score: 0; Maximum score: 54 Higher score = higher engagement at work (better outcome)
Urine oxytocin | Two samples were taken one hour apart at baseline, and this was repeated three months later.
  Change from baseline in the level of urine oxytocin before and after each intervention. This is an exploratory study so the maximum and minimum values are not known, and any change up or down is interesting.
Salivary Oxytocin | Two samples were taken one hour apart at baseline, and this was repeated three months later
  Change from baseline in the level of salivary oxytocin before and after each intervention. This is an exploratory study so the maximum and minimum values are not known, and any change up or down is interesting.
Salivary Cortisol | Two samples were taken one hour apart at baseline, and this was repeated three months later
  Change from baseline in the level of salivary cortisol before and after each intervention. This is an exploratory study so the maximum and minimum values are not known, and any change up or down is interesting.
Hair Cortisol | Change over the three month study period. Baseline measurement and immediately after final intervention.
  Change from baseline in hair cortisol levels. Maximum and minimum levels are not known and any change up or down is interesting.
Work Empowerment Scale | Change over the three month study period. Baseline measurement and immediately after final intervention.
  Minimum score: 12; Maximum score: 84 Change from baseline on Work Empowerment Scale before and after intervention. Higher score = higher empowerment at work (better outcome)

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No